CLINICAL TRIAL: NCT06544369
Title: Prospective Study on COVID -19 Reinfection on Vaccinated and Non-vaccinated Outpatients
Status: Completed | Type: Observational
Sponsor: Soad Ali (Other)
Responsible Party: Sponsor-Investigator, Soad Ali, lecturer of pharmaceutics and clinical pharmacy Deraya university, Deraya University
Organization: Deraya University (Other)
Other Study IDs: Deraya university
Record Dates: First submitted 2021-10-25; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccinated group: all criteria are accepted for study
  Interventions: Biological: COVID-19 vaccin
- Non-vaccinated group: all criteria are accepted for study
  Interventions: Biological: COVID-19 vaccin

INTERVENTIONS:
Biological: COVID-19 vaccin — injection

SUMMARY:
the aim of the study is to compare the severity of symptoms in case of reinfection with COVID-19. the study will compare between two groups; vaccinated and non vaccinated. the side effects from vaccination and symptoms of infection and reinfection will be reprted.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with COVID infection
* take any type of vaccines

Exclusion Criteria:

* no accept sharing
* not vaccinated with COVID vaccine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the study group are infected patients with COVID-19
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
percent of reinfection with COVID-19 in vaccinated and non vaccinated | one year

SECONDARY OUTCOMES:
scoring of symptoms in case of reinfection in vaccinated and non vaccinated | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Minya, Egypt